CLINICAL TRIAL: NCT03665038
Title: A Multicenter, Open-Label Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Brexanolone in the Treatment of Adolescent Female Subjects With Postpartum Depression
Brief Title: A Study to Assess the Safety of Brexanolone in the Treatment of Adolescent Female Participants With Postpartum Depression (PPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 547-PPD-304; 2017-004356-34 (EudraCT Number)
Record Dates: First submitted 2018-04-30; First posted 2018-09-11 (Actual); Results first posted 2022-08-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2022-07

CONDITIONS: Post Partum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — brexanolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brexanolone (Experimental): Participants will receive a 60-hour single continuous IV infusion of brexanolone, at 30 mcg/kg/hour (0 to 4 hours), at 60 mcg/kg/hour (4 to 24 hours), at 90 mcg/kg/hour (24 to 52 hours), followed by a taper to 60 mcg/kg/hour (52 to 56 hours), and 30 mcg/kg/hour (56 to 60 hours) during the study.
  Interventions: Drug: Brexanolone

INTERVENTIONS:
Drug: Brexanolone — Administered as IV infusion.

SUMMARY:
This is a multi-center study evaluating the safety, tolerability, and pharmacokinetics of brexanolone in the treatment of adolescent female participants with postpartum depression (PPD).

ELIGIBILITY:
Key Inclusion Criteria:

1. Participant has had a major depressive episode that began no earlier than the third trimester and no later than the first 4 weeks following delivery, as diagnosed by Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) Axis I Disorders (SCID-5).
2. Participant is ≤6 months postpartum at screening.

Key Exclusion Criteria:

1. Active psychosis
2. Attempted suicide during current episode of PPD
3. Medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder.

Note: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 15 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Sage Investigational Site, Tempe, Arizona
  - Sage Investigational Site, North Little Rock, Arkansas
  - Sage Investigational Site, Miramar, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Pensacola, Florida
  - Sage Investigational Site, Pinellas Park, Florida
  - Sage Investigational Site, Pompano Beach, Florida
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Decatur, Georgia
  - Sage Investigational Site, Edgewood, Kentucky
  - Sage Investigational Site, Owensboro, Kentucky
  - Sage Investigational Site, Flowood, Mississippi
  - Sage Investigational Site, Jackson, Mississippi
  - Sage Investigational Site, Chapel Hill, North Carolina
  - Sage Investigational Site, Middleburg Heights, Ohio
  - Sage Investigational Site, Houston, Texas
  - Sage Investigational Site, League City, Texas

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

REFERENCES:
- See also: Related Info — http://www.sagerx.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigating sites in the United States, from 07 September 2018 to 08 January 2021.
Pre-assignment Details: As per Protocol Versions 1 through 3, the study was initiated as a double-blind, placebo-controlled study, in which participants received brexanolone or brexanolone-matching placebo in a blinded manner. As per Protocol Version 4, the study was transitioned to an open-label study, where all participants received brexanolone.
Groups:
- Double-Blind Phase: Placebo: Participants received a 60-hour single continuous intravenous (IV) infusion of brexanolone-matching placebo, at 30 micrograms per kilogram per hour (mcg/kg/hour) (0 to 4 hours), at 60 mcg/kg/hour (4 to 24 hours), at 90 mcg/kg/hour (24 to 52 hours), followed by a taper to 60 mcg/kg/hour (52 to 56 hours), and 30 mcg/kg/hour (56 to 60 hours) during double-blind phase of the study.
- Double-Blind Phase: Brexanolone: Participants received a 60-hour single continuous IV infusion of brexanolone, at 30 mcg/kg/hour (0 to 4 hours), at 60 mcg/kg/hour (4 to 24 hours), at 90 mcg/kg/hour (24 to 52 hours), followed by a taper to 60 mcg/kg/hour (52 to 56 hours), and 30 mcg/kg/hour (56 to 60 hours) during double-blind phase of the study.
- Open-Label Phase: Brexanolone: Participants received a 60-hour single continuous IV infusion of brexanolone, at 30 mcg/kg/hour (0 to 4 hours), at 60 mcg/kg/hour (4 to 24 hours), at 90 mcg/kg/hour (24 to 52 hours), followed by a taper to 60 mcg/kg/hour (52 to 56 hours), and 30 mcg/kg/hour (56 to 60 hours) during open-label phase of the study.
Period: Overall Study
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: Brexanolone | Open-Label Phase: Brexanolone
Started | 8 | 8 | 12
Completed | 8 | 8 | 11
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety set included all participants administered study drug.
Groups:
- Double-Blind Phase: Placebo: Participants received a 60-hour single continuous IV infusion of brexanolone-matching placebo, at 30 mcg/kg/hour (0 to 4 hours), at 60 mcg/kg/hour (4 to 24 hours), at 90 mcg/kg/hour (24 to 52 hours), followed by a taper to 60 mcg/kg/hour (52 to 56 hours), and 30 mcg/kg/hour (56 to 60 hours) during double-blind phase of the study.
- Total: Total of all reporting groups
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: Brexanolone | Open-Label Phase: Brexanolone | Total
Number analyzed (Participants) | 8 | 8 | 12 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.6 (0.52) | 16.4 (0.52) | 16.3 (0.78) | 16.4 (0.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 12 | 28
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 8 | 6 | 12 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 10 | 22
  White | 2 | 2 | 1 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is defined as an AE with onset on or after the start of study drug infusion, or any worsening of a pre-existing medical condition/AE with onset on or after the start of study drug infusion.
Time Frame: From first dose of study drug up to end of follow-up period (up to Day 30)
Population: The safety set included all participants administered study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: Brexanolone | Open-Label Phase: Brexanolone
Number analyzed (Participants) | 8 | 8 | 12
Participants | 4 | 3 | 5

2. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) From Time Zero to 60 Hours (AUC0-60)
Time Frame: Day 1: From 0 hour (pre-infusion) and at 4, 8, 12, 24, 30, 36, 48 hours during the infusion; at 60 hours (end of infusion)
Population: The pharmacokinetic (PK) set included participants in the safety set for whom at least one evaluable post-baseline PK sample with a measurable brexanolone concentration was available.
Measure: Mean (Standard Deviation); unit: hours*nanograms per milliliter(hr*ng/mL)
Arm/Group | Double-Blind Phase: Brexanolone | Open-Label Phase: Brexanolone
Number analyzed (Participants) | 8 | 11
hours*nanograms per milliliter(hr*ng/mL) | 3694.9 (397.90) | 3516.0 (562.85)

3. Secondary Outcome: AUC From Time Zero to Infinity (AUCinf)
Time Frame: as for outcome 2
Population: The PK set included participants in the safety set for whom at least one evaluable post-baseline PK sample with a measurable brexanolone concentration was available.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Double-Blind Phase: Brexanolone | Open-Label Phase: Brexanolone
Number analyzed (Participants) | 8 | 11
hr*ng/mL | 4125.9 (481.84) | 3982.2 (709.70)

4. Secondary Outcome: Maximum (Peak) Plasma Concentration (Cmax)
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Double-Blind Phase: Brexanolone | Open-Label Phase: Brexanolone
Number analyzed (Participants) | 8 | 11
nanograms per milliliter (ng/mL) | 85.31 (9.571) | 81.66 (13.528)

5. Secondary Outcome: Time at Maximum (Peak) Plasma Concentration (Tmax)
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Double-Blind Phase: Brexanolone | Open-Label Phase: Brexanolone
Number analyzed (Participants) | 8 | 11
hour (hr) | 52.20 [52.0 to 52.4] | 52.30 [52.1 to 54.9]

6. Secondary Outcome: Steady-State Drug Concentration in the Plasma During Constant-Rate Infusion (Css)
Description: Given that brexanolone is infused to steady-state plasma concentrations, the model-predicted steady-state drug concentration in the plasma during constant-rate infusion value also represents the predicted maximum plasma concentration at the highest infused dose (90 ug/kg/h).
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Number; unit: ng/mL
Arm/Group | Double-Blind Phase: Brexanolone | Open-Label Phase: Brexanolone
Number analyzed (Participants) | 8 | 11
ng/mL | 79.4 | 79.4

7. Secondary Outcome: Average Drug Concentration in Plasma at Steady State During a Dosing Interval (Cavg)
Description: Cavg was evaluated as the time-weighted average plasma concentrations of brexanolone over the interval.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Double-Blind Phase: Brexanolone | Open-Label Phase: Brexanolone
Number analyzed (Participants) | 8 | 11
ng/mL | 61.59 (6.639) | 58.60 (9.386)

8. Secondary Outcome: Half-Life of First Elimination Phase of Brexanolone (Thalf)
Description: Half-life is the time required for half of the drug to be eliminated from the serum.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Double-Blind Phase: Brexanolone | Open-Label Phase: Brexanolone
Number analyzed (Participants) | 8 | 11
hour | 12.24 (0.466) | 12.55 (1.096)

9. Secondary Outcome: Clearance of Brexanolone (CL/F)
Description: Clearance is defined as the volume of plasma from which a substance is completely removed per unit time.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: liters per hour (L/hr)
Arm/Group | Double-Blind Phase: Brexanolone | Open-Label Phase: Brexanolone
Number analyzed (Participants) | 8 | 11
liters per hour (L/hr) | 66.86 (13.858) | 77.88 (18.026)

10. Secondary Outcome: Steady-State of Volume of Distribution (Vss)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: liters (L)
Arm/Group | Double-Blind Phase: Brexanolone | Open-Label Phase: Brexanolone
Number analyzed (Participants) | 8 | 11
liters (L) | 448.1 (70.34) | 588.5 (187.53)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of follow-up period (up to Day 30)
Description: The safety set included all participants administered study drug.
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: Brexanolone | Open-Label Phase: Brexanolone
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 1/12
Other Adverse Events (participants affected / at risk) | 4/8 | 3/8 | 4/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Phase: Placebo (N=8) | Double-Blind Phase: Brexanolone (N=8) | Open-Label Phase: Brexanolone (N=12)
Dizziness (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Phase: Placebo (N=8) | Double-Blind Phase: Brexanolone (N=8) | Open-Label Phase: Brexanolone (N=12)
Dizziness (Nervous system disorders) | 0 | 0 | 2
Sedation (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Infusion site pain (General disorders) | 0 | 2 | 1
Infusion site extravasation (General disorders) | 1 | 0 | 0
Infusion site inflammation (General disorders) | 1 | 0 | 0
Infusion site swelling (General disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1
Localized infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT03665038/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT03665038/SAP_001.pdf